CLINICAL TRIAL: NCT02360683
Title: Predictive Factors for Therapeutic Response of Subthalamic Stimulation on Quality of Live in Parkinson's Disease
Brief Title: Predictive Factors and Subthalamic Stimulation in Parkinson's Disease
Acronym: PREDI-STIM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011_41; 2013-A00193-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-01-05; First posted 2015-02-10 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Parkinson's Disease
Keywords: Subthalamic neurostimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Parkinson's disease: Large population of Parkinson's patients who benefit from subthalamic stimulation
  Interventions: Other: patients with Parkinson's disease

INTERVENTIONS:
Other: patients with Parkinson's disease
  Other Names: systematic and standardized collection of data

SUMMARY:
This study identify preoperative predictors of response to subthalamic stimulation at 1 year, 3 years and 5 years in terms of quality of life, from a broad prospective multicenter study French with standardized collection of clinical data , imaging and genetic .

The investigators want to identify factors that predict the improvement of quality of life for one year corresponding to a decrease of PDQ39 score of at least 20 %. They believe that improvement would be less likely to become zero to 3 or 5 years and question the indication of the subthalamic stimulation (risks and costs). This is part of a process of "personalization" of the therapeutic care that is of any interest to the subthalamic stimulation. It is a therapeutic option that could be dangerous if patient selection is not optimal , and expensive, if the benefit is not large enough to reduce the number of medications and hospitalizations medium term . In addition, it will quantify the improvement of quality of life in the longer term and harmonize national assessments .

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a pre- therapeutic assessment and therapeutic monitoring for one year , 3 years and 5 years as part of the regular monitoring of the subthalamic stimulation
* Bilateral STN stimulation considered
* Patient able to provide their free and informed consent
* Patient with insurance coverage

Exclusion Criteria:

* Atypical Parkinson's disease do not meet the criteria of stuff .
* MP under 5 years
* Severe cognitive impairment or dementia ( Score Moca <24 and DSM-IV criteria)
* Parkinson's Psychosis
* Reply to L- dopa <30 %
* Against indication for surgery
* Severe brain atrophy or abnormal MRI
* The presence of another very serious condition terminal life- short-term prognosis ( malignancy ) is an indication against .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric French cohort of 1000 Parkinson's disease patients, for obtain 400 patients in the failure group
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Improve of quality of life on PDQ39>20% | 1 year

SECONDARY OUTCOMES:
Percentage of motor score MDS-UPDRS III improve under stimulation | 1 year
Socio-familial evolution (institutionalization) | 1, 3 and 5 years
Clinical Global Impression of Patient by 7-point scale | 1, 3 and 5 years
  with the CGI-scale
Clinical Global Impression of doctor by 7-point scale | 1, 3 and 5 years
  with the CGI-scale
Death | 1, 3 and 5 years
Cognitive function with a neuropsychological examination | 1, 3 and 5 years
  with Mattis scale, Wisconsin Card Sorting test, Stroop test, , verbal episodic memory test with 16 items, phonemic and semantic verbal fluency, Boston naming test (15 items), clock drawing and Benton line orientation task
Behavior test | 1, 3 and 5 years
  ECMP scale of Ardouin 2009, Hamilton depression scale, Anxiety Hamilton scale, Lille Apathy Rating Scale, QUIP questionnaire, Billieux Impulsivity Scale, Hallucination questionnaire of Miami
Motor response rates to Levodopa | 1, 3 and 5 years
  with the difference of the motor handicap measured by MDS UPDRS part III before and after an acute L-dopa challenge
Non-motor functions evaluated by a numerical evaluation scale | screening and at 1, 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David DEVOS, MD, PhD, Study Chair — University Hospital, Lille
Locations (15):
- France (15):
  - CHU Hôpital NORD, Amiens
  - Hôpital Pierre Wertheimer, Bron
  - Chu Gabriel-Montpied, Clermont-Ferrand
  - Devos, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Central,, Nancy
  - CHU hôpital Nord Laennec, Nantes
  - Hôpital Pasteur, Nice
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hopital Pitie Salpetriere, Paris
  - CHU de Poitiers, Poitiers
  - CHU Hôpital Pontchaillou, Rennes
  - Chu Ch.Nicolle, Rouen
  - Hôpital de Hautepierre, Strasbourg
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ollivier T, Pinto S, Rolland AS, Cailliau E, Touzet G, Thobois S, Eusebio A, Hainque E, Rouaud T, Drapier S, Guehl D, Maltete D, Anheim M, Lagha Boukbiza O, Giordana C, Tir M, Hopes L, Hubsch C, Jarraya B, Marques A, Brefel C, Rascol O, Corvol JC, Benatru I, Defebvre L, Devos D, Moreau C; French PREDISTIM study group. Parkinson's Disease, Speech and Neurosurgery. Brain Behav. 2025 May;15(5):e70101. doi: 10.1002/brb3.70101. PMID 40302158
- [Derived] Meyer M, Spitz E, Colnat-Coulbois S, Benatru I, Guehl D, Hainque E, Rolland AS, Corvol JC, Devilliers H, Schwan R, Devos D; PREDISTIM group. Development and validation of the DBS-PS (Deep Brain Stimulation-Perception Scale): Assessing parkinsonian patients' expectations to prevent post-operative disappointment? J Neurol Sci. 2024 Jul 15;462:123093. doi: 10.1016/j.jns.2024.123093. Epub 2024 Jun 13. PMID 38908172
- [Derived] Rolland AS, Touzet G, Carriere N, Mutez E, Kreisler A, Simonin C, Kuchcinski G, Chalhoub N, Pruvo JP, Defebvre L, Reyns N, Devos D, Moreau C. The Use of Image Guided Programming to Improve Deep Brain Stimulation Workflows with Directional Leads in Parkinson's Disease. J Parkinsons Dis. 2024;14(1):111-119. doi: 10.3233/JPD-225126. PMID 38189764
- [Derived] Boussac M, Arbus C, Colin O, Laurencin C, Eusebio A, Hainque E, Corvol JC, Versace N, Rascol O, Rousseau V, Harroch E, Ory-Magne F, Fabbri M, Moreau C, Rolland AS, Jarraya B, Maltete D, Drapier S, Marques AR, Auzou N, Wirth T, Meyer M, Giordana B, Tir M, Rouaud T, Devos D, Brefel-Courbon C; PREDISTIM study group. Personality assessment with Temperament and Character Inventory in Parkinson's disease. Parkinsonism Relat Disord. 2022 Oct;103:34-41. doi: 10.1016/j.parkreldis.2022.08.004. Epub 2022 Aug 19. PMID 36030666
- [Derived] Besse-Pinot E, Pereira B, Durif F, Fantini ML, Durand E, Debilly B, Derost P, Moreau C, Hainque E, Rouaud T, Eusebio A, Benatru I, Drapier S, Guehl D, Rascol O, Maltete D, Lagha-Boukbiza O, Giordana C, Tir M, Thobois S, Hopes L, Hubsch C, Jarraya B, Rolland AS, Corvol JC, Devos D, Marques A; Predistim Study Group. Preoperative REM Sleep Behavior Disorder and Subthalamic Nucleus Deep Brain Stimulation Outcome in Parkinson Disease 1 Year After Surgery. Neurology. 2021 Nov 16;97(20):e1994-e2006. doi: 10.1212/WNL.0000000000012862. Epub 2021 Oct 19. PMID 34667082
- [Derived] Betrouni N, Moreau C, Rolland AS, Carriere N, Chupin M, Kuchcinski G, Lopes R, Viard R, Defebvre L, Devos D. Texture-based markers from structural imaging correlate with motor handicap in Parkinson's disease. Sci Rep. 2021 Feb 1;11(1):2724. doi: 10.1038/s41598-021-81209-4. PMID 33526820
- [Derived] Boussac M, Arbus C, Dupouy J, Harroch E, Rousseau V, Croiset A, Ory-Magne F, Rascol O, Moreau C, Rolland AS, Maltete D, Rouaud T, Meyer M, Drapier S, Giordana B, Anheim M, Hainque E, Jarraya B, Benatru I, Auzou N, Belamri L, Tir M, Marques AR, Thobois S, Eusebio A, Corvol JC, Devos D, Brefel-Courbon C; PREDI-STIM study group. Personality dimensions of patients can change during the course of parkinson's disease. PLoS One. 2021 Jan 7;16(1):e0245142. doi: 10.1371/journal.pone.0245142. eCollection 2021. PMID 33411732
- [Derived] Santin MDN, Voulleminot P, Vrillon A, Hainque E, Bereau M, Lagha-Boukbiza O, Wirth T, Montaut S, Bardinet E, Kyheng M, Rolland AS, Voirin J, Drapier S, Durif F, Eusebio A, Giordana C, Auzou N, Houeto JL, Hubsch C, Jarraya B, Laurencin C, Maltete D, Meyer M, Rascol O, Rouaud T, Tir M, Moreau C, Corvol JC, Proust F, Grabli D, Devos D, Tranchant C, Anheim M; Predistim Study Group. Impact of Subthalamic Deep Brain Stimulation on Impulse Control Disorders in Parkinson's Disease: A Prospective Study. Mov Disord. 2021 Mar;36(3):750-757. doi: 10.1002/mds.28320. Epub 2020 Oct 6. PMID 33022101
- [Derived] Boussac M, Arbus C, Dupouy J, Harroch E, Rousseau V, Ory-Magne F, Rascol O, Moreau C, Maltete D, Rouaud T, Meyer M, Houvenaghel JF, Marse C, Tranchant C, Hainque E, Jarraya B, Ansquer S, Bonnet M, Belamri L, Tir M, Marques AR, Danaila T, Eusebio A, Devos D, Brefel-Courbon C; PREDI-STIM study group*. Personality Dimensions Are Associated with Quality of Life in Fluctuating Parkinson's Disease Patients (PSYCHO-STIM). J Parkinsons Dis. 2020;10(3):1057-1066. doi: 10.3233/JPD-191903. PMID 32444557